CLINICAL TRIAL: NCT01413191
Title: Phase II Study of IMC-A12 in Metastatic Uveal Melanoma
Brief Title: Cixutumumab in Treating Patients With Metastatic Melanoma of the Eye
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02228; NCI-2011-02228 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2010-0451 (Other: M D Anderson Cancer Center); 8832 (Other: CTEP); P30CA016672 (NIH); N01CM00039 (NIH)
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Results first posted 2015-07-20 (Estimated); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Ciliary Body and Choroid Melanoma, Medium/Large Size; Ciliary Body and Choroid Melanoma, Small Size; Iris Melanoma; Metastatic Intraocular Melanoma; Recurrent Intraocular Melanoma; Stage IV Intraocular Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — cixutumumab

ARMS (1):
- CixutumumabTreatment (Experimental): Cixutumumab 10 mg/kg intravenous (IV) over 1 hour on days 1 and 15 for 4 week courses.
  Interventions: Biological: Cixutumumab; Other: Laboratory biomarker analysis

INTERVENTIONS:
Biological: Cixutumumab — 10 mg/kg IV infusion over 1 hour every 2 weeks with treatment cycle defined as 4 weeks
  Other Names: anti-IGF-1R recombinant monoclonal antibody IMC-A12; IMC-A12
Other: Laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving cixutumumab works in treating patients with metastatic melanoma of the eye. Monoclonal antibodies, such as cixutumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate of metastatic uveal melanoma when treated with IMC-A12 (cixutumumab).

II. To determine the safety and tolerability of IMC-A12 in patients with metastatic uveal melanoma.

SECONDARY OBJECTIVES:

I. To determine the disease control rate of patients treated with IMC-A12. II. To determine the duration of response of patients treated with IMC-A12. III. To determine the progression-free survival and overall survival of patients treated with IMC-A12.

TERTIARY OBJECTIVES:

I. To correlate the presence of GNAQ and GNA11 mutations with response to IMC-A12.

II. To correlate the expression of IGF-1R with response to IMC-A12. III. To determine the effect of IMC-A12 on expression of proteins involved in initiation, growth, and spread of uveal melanoma cells.

IV. To determine resistance mechanisms to IMC-A12.

OUTLINE: This is a multicenter study.

Patients receive cixutumumab intravenously (IV) over 1 hour on days 1 and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Archived and fresh tumor tissue and serum samples may be collected for correlative studies.

After completion of study treatment, patients are followed up for 30 days and then every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a history of uveal melanoma and documented metastatic disease
* Patients must have at least one unidimensionally measurable lesion; if this is a cutaneous lesion it must be at least 10 mm by caliper measure; if it is a visceral or nodal or soft tissue lesion, it must be clearly measurable > 20 mm with conventional techniques or > 10 mm with spiral CT scan; bone lesions are not considered measurable
* One prior systemic chemotherapy and any number of immunotherapies or vaccine therapies are allowed; prior treatment with hepatic arterial chemotherapy infusion or perfusion or chemoembolization of liver metastasis is allowed; prior treatment with radiation therapy is allowed but not more than 3000 cGy to fields including substantial marrow; patients are not required to have had prior therapy

  * At least 6 weeks (42 days) since any prior immunotherapy, cytokine, biologic, vaccine or other therapy unless patients have progressed during therapy; if progression occurred during therapy, patient must have recovered from any side effects
  * At least 4 weeks (28 days) since prior radiotherapy and prior adjuvant chemotherapy
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2
* Patients must have a life expectancy of at least 3 months
* Leukocytes > 3,000/mm3
* Absolute neutrophil count ≥ 1,500/mm3
* Hemoglobin ≥ 9.0 g/dL
* Platelets ≥ 100,000/mm3
* Aspartate transaminase-alanine transaminase ratio (AST(SGOT)/ALT(SGPT)) ≤ 3 times institutional upper limit of normal (ULN); ≤ 5 times institutional ULN if liver metastases present
* Total bilirubin < 1.5 times institutional ULN
* Creatinine < 1.5 times institutional ULN OR creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Fasting serum glucose < 120 mg/dL or < institutional ULN
* Patients must have no angina at rest
* The effects of IMC-A12 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because monoclonal antibodies could be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and for 3 months after the last dose of IMC-A12; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Both men and women and members of all races and ethnic groups are eligible for this trial
* Patients must have the ability to understand and the willingness to sign a written informed consent form indicating that they are aware of the investigational nature of this study and in keeping with the policies of the institution

Exclusion Criteria:

* Patients whose site of primary melanoma is not uveal
* Patients who have a current history of neoplasm other than the entry diagnosis except for curatively treated non-melanoma skin cancer or carcinoma in situ of the cervix or other cancers treated for cure and with a disease-free survival longer than 5 years
* Patients with symptomatic central nervous system metastasis including those with central nervous system (CNS) metastasis who require oral steroids for cerebral edema or have progression on CT/MRI
* Patients who are pregnant or nursing and patients who are not practicing an acceptable method of birth control; patients may not breast-feed while on this study; pregnant women are excluded from this study because IMC-A12 is a monoclonal antibody with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IMC-A12, breastfeeding women are excluded
* Patients with current active infections requiring anti-infectious treatment (e.g., antibiotics, antivirals, or antifungals)
* Patients with poorly controlled diabetes mellitus; patients with a history of diabetes mellitus are allowed to participate, provided that their blood glucose is within normal range (fasting < 120 mg/dL or below institutional ULN) and that they are on a stable dietary or therapeutic regimen for this condition
* Patients with unstable or serious concurrent medical conditions are excluded; examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Patients with one or more of the following as the only manifestations of disease are ineligible: leptomeningeal disease, ascites, pleural/pericardial effusions, carcinomatous lymphangitis
* Patients with Gilbert's Syndrome
* Patients must not have had major surgery within the past 14 days
* Patients must not receive any concurrent chemotherapy or immunotherapy while on study; only palliative radiotherapy is permitted to symptomatic lesions in which event the irradiated lesions may not be considered target or non-target lesions for response; palliative radiation immediately before or during the study is acceptable provided there is evaluable disease that has been radiated; palliative radiation is acceptable provided that the irradiated lesions are not used to determine response assessment
* HIV-positive patients with an absolute CD4 count < 300 K/uL
* Patients may not be receiving any other investigational agents
* Patients with a history of treatment with other agents targeting the insulin-like growth factor pathway
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to IMC-A12

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-08; Primary Completion 2013-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Patel, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 02, 2011 to August 23, 2012. Recruitment was done at The University of Texas MD Anderson Cancer Center (MD Anderson) and The Thomas Jefferson University.
Period: Overall Study
Arm/Group | CixutumumabTreatment
Started | 18
Completed | 7
Not Completed | 11
Not completed — Lost to Follow-up | 5
Not completed — Disease Progression | 5
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 67 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: Response rate is the percentage of subjects with a confirmed complete or partial response using revised Response Evaluation Criteria in Solid Tumors (RECIST) where changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria: Complete Response (CR): Disappearance all target lesions; pathological lymph nodes reduction in short axis to <10 mm. Partial Response (PR): 30% or > decrease in sum diameters of target lesions, reference baseline sum diameters. Progressive Disease (PD): 20% or > increase in sum diameters of target lesions, reference smallest sum on study (includes baseline sum if smallest on study); and sum must demonstrate absolute increase of 5+ mm. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, reference smallest sum diameters while on study.
Time Frame: Baseline to 2 years
Population: One participant was not evaluable for response assessment.
Measure: Number; unit: participants
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 17
participants
  CR | 0
  PR | 0
  PD | 8
  SD | 9

2. Secondary Outcome: Disease Control Rate
Description: Disease Control Rate is the proportion of subjects with a confirmed complete or partial response of any duration or stable disease ≥3 months in duration.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 18
Participants
  PR | 0
  CR | 0
  SD | 9

3. Secondary Outcome: Duration of Response
Description: Duration of response will be summarized by using descriptive statistics. Median duration of response will be estimated by using the Kaplan-Meier method.
Time Frame: From the date criteria are first met for complete or partial response until the first date of documented progression, assessed up to 2 years
Population: Duration of response could not be calculated, as there were no responders.
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: WEEKS
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 18
WEEKS | 12.21 [0 to 23.2]

5. Secondary Outcome: Overall Survival (OS)
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: WEEKS
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 18
WEEKS | 59.71 [0 to 109.6]

6. Secondary Outcome: Durable Response Rate
Description: Durable Response Rate is the proportion of subjects with a confirmed complete or partial response ≥ 6 months in duration.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 17
Participants | 0

7. Other Pre Specified Outcome: Tumor Shrinkage for All Efficacy-evaluable Patients
Time Frame: Up to 2 years
Population: No participants was evaluable due to progression.
Arm/Group | CixutumumabTreatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events reporting includes occurrences within 30 days of the last investigational agent/intervention. Overall study period: August 2011 to May 2014.
Arm/Group | CixutumumabTreatment
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CixutumumabTreatment (N=18)
Dehydration (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CixutumumabTreatment (N=18)
Abdominal pain (Gastrointestinal disorders) | 9 (14)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 2 (4)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 3 (3)
Allergic rhinitis (Immune system disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 10 (15)
Anorexia (Gastrointestinal disorders) | 11 (13)
Anxiety (Nervous system disorders) | 1 (1)
Arthralgia (Cardiac disorders) | 2 (2)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 8 (9)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Blood bilirubin increased (Metabolism and nutrition disorders) | 3 (3)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Chest wall pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholesterol high (Metabolism and nutrition disorders) | 8 (15)
Confusion (Nervous system disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 7 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Gastrointestinal disorders) | 2 (2)
Depression (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (19)
Dizziness (Nervous system disorders) | 5 (7)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (7)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Gastrointestinal disorders) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear and labyrinth disorders, Other (Ear and labyrinth disorders) | 4 (4)
Edema limbs (Musculoskeletal and connective tissue disorders) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Eye disorders, Other (Eye disorders) | 2 (2)
Eye pain (Eye disorders) | 2 (2)
Fatigue (General disorders) | 17 (26)
Floaters (Eye disorders) | 9 (9)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - (Other) (Gastrointestinal disorders) | 1 (1)
Pain NOS (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Glucose intolerance (Endocrine disorders) | 1 (1)
Headache (Nervous system disorders) | 4 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (29)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypertension (Cardiac disorders) | 12 (45)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 9 (20)
Hyperuricemia (Metabolism and nutrition disorders) | 5 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Cardiac disorders) | 2 (3)
Hypothermia (General disorders) | 2 (4)
Infections and infestations - (Other) (Infections and infestations) | 3 (4)
Investigations - (Other) (Investigations) | 1 (1)
Lethargy (General disorders) | 1 (1)
Lipase increased (Metabolism and nutrition disorders) | 6 (7)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (3)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (20)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - (Other) (Nervous system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 2 (3)
Pain (General disorders) | 7 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (6)
Pancreatitis (Hepatobiliary disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 5 (5)
Penile infection (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Platelet count decreased (Blood and lymphatic system disorders) | 7 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (8)
Psychiatric disorders - (Other) (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Respiratory, thoracic and mediastinal disorders - (Other) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Serum amylase increased (Metabolism and nutrition disorders) | 3 (8)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Skin and subcutaneous tissue disorders - (Other) (Skin and subcutaneous tissue disorders) | 3 (3)
Somnolence (Nervous system disorders) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (6)
Weight loss (General disorders) | 8 (14)
White blood cell decreased (Blood and lymphatic system disorders) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less